CLINICAL TRIAL: NCT05124834
Title: Evaluierung Der Systemgenauigkeit Des JT100 Blood Glucose Monitoring Systems Der Firma Tyson Bioresearch Inc. gemäß DIN EN ISO 15197:2015
Brief Title: System Accuracy of the Blood Glucose Monitor for Personal Use JT100
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Collaborators: Tyson Bioresearch Inc., Kedong 3rd Rd., Zhunan Township, Miaoli County 35053, Taiwan (Unknown)
Responsible Party: Principal Investigator, Matthes Kenning, Dr. Eckhard Salzsieder, Director, Institut fur Diabetes Karlsburg GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDK_ISO_2021_004
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject glucometer measurement (Experimental): Blood glucose measurement BGM for personal use
  Interventions: Diagnostic Test: blood glucose measurement, blood glucose monitor for personal use; Diagnostic Test: blood glucose measurement, laboratory reference device

INTERVENTIONS:
Diagnostic Test: blood glucose measurement, blood glucose monitor for personal use — measurement of the blood glucose concentration using the blood glucose monitor for personal use (TJ100)
  Other Names: measurement of the blood glucose concentration using the blood glucose monitor for personal use (TJ100)
Diagnostic Test: blood glucose measurement, laboratory reference device — measurement of the blood glucose concentration using a laboratory reference device (YSI 2300 Stat Plus)

SUMMARY:
This study assesses the system accuracy a blood glucose monitoring systems pursuant to ISO 15197

DETAILED DESCRIPTION:
This study assesses the system accuracy the blood glucose monitoring systems for personal use TJ100 pursuant to ISO 15197:2015 guidelines

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with clinical indication for blood glucose testing
* Signed form of consent
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study

Exclusion Criteria:

* Pregnancy or lactation
* Severe acute disease (at study physician's discretion)
* Acute or chronic diseases with inherent risk of aggravation by the procedure (at study physician's discretion)
* Current constitution that does not allow participating in the study (e.g. hematocrit out of
* the devices's specifications, medication known to influence blood glucose measurements; Appendix A of ISO 15197)
* Being unable to give informed consent
* Age younger than 18 years
* Legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | day 1
  Assessment of the analytical measurement performance of the blood glucose monitor based on procedures defined in DIN EN ISO 15197

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Salzsieder, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No